CLINICAL TRIAL: NCT03458949
Title: Pilot Study in a Company in Maine-et-Loire to Evaluate the Feasibility, Acceptability, and Impact on the Participation Rate of Awareness of Colorectal Cancer Screening by Occupational Health Teams
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DETECT
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: awareness campaign — awareness campaign for colorectal cancer screening in the workplace

SUMMARY:
The main objective of this pilot study is to implement an awareness campaign for colorectal cancer screening in the workplace, in partnership with the staff of the occupational health service of one of the largest companies in Maine-Loire , and to evaluate the impact of this action on the participation rate of colorectal cancer screening among employees.

ELIGIBILITY:
Inclusion Criteria:

* The study population is made up of the employees of the CHU d'Angers included in the target population of organized colorectal cancer screening in the Maine-et-Loire so employees aged 50 and over.

Exclusion Criteria:

* The criteria for non-inclusion are those of organized screening for colorectal cancer taking into account the active population:
* Age <50 years and> 67 years
* Personal or family history of polyps or colorectal cancer
* Personal history of intestinal disease already undergoing colonoscopy surveillance (chronic inflammatory bowel disease, HNPCC syndrome, familial adenomatous polyposis)
* Known genetic disease with risk of developing colorectal cancer.

Ages: 50 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
variation of the rate of participation in colorectal cancer screening | 2 years
  effective variation (after versus prior to awareness raising) of the overall rate of participation in colorectal cancer screening among employees of the company after 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: François-Xavier Caroli-Bosc, MDPhD, Principal Investigator — University Hospital, Angers
Locations (1):
- Santé au Travail CHU Angers, Angers, France